CLINICAL TRIAL: NCT03616327
Title: Workflow Validation of an In-Home Feedback Controlled Mandibular Positioner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zephyr Sleep Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZCP201705
Record Dates: First submitted 2018-01-08; First posted 2018-08-06 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MATRx in-lab or MATRx plus test (Other): Participants will undergo the MATRx in-lab or MATRx plus home test to determine adequacy for mandibular repositioning oral appliance therapy. The tests only differ in their setting (i.e., in the sleep lab or at home). All participants will receive the same treatment protocol preceding and following the MATRx/MATRx plus test.
  Interventions: Device: MATRx in-lab, MATRx plus

INTERVENTIONS:
Device: MATRx in-lab, MATRx plus — The MATRx remotely controlled mandibular positioner (RCMP) consists of temporary dental trays connected to an extra-oral linear actuator that protrudes the mandible. MATRx is used during polysomnography, where sleep and cardio-respiratory variables are recorded during sleep. The position of the mandible is controlled remotely by a sleep technologist, who moves the mandible while monitoring cardio-respiratory variables. The test determines if mandibular protrusion eliminates pharyngeal obstruction and the required protrusion. The MATRx plus is used in the home. Like the RCMP, the patient sleeps with the motorized mandibular positioner (MP) in place. However, the MP's position is controlled by a computer, making it a feedback controlled mandibular positioner (FCMP). The FCMP detects apneas and hypopneas in real time. Using this information, the controller decides when to move the mandible and by how much. The test predicts of therapeutic outcome with OA and provides a target protrusion.

SUMMARY:
The purpose of the study is to test the workflow of the MATRx and MATRx plus feedback controlled mandibular positioner in its intended setting and considerations related to decision making by the care provider. The workflow includes the participant's recruitment into the study, the screening process, visits at the dentist, home sleep tests, and the decision made regarding oral appliance therapy based on the results of the sleep tests.

DETAILED DESCRIPTION:
Sleep apnea (OSA) is a condition in which the air passage in the throat closes or partly closes during sleep and repeatedly interrupts breathing. The standard treatment of sleep apnea is continuous positive airway pressure (CPAP) applied to the nose, but it is not suitable for all patients. Another treatment is to use an oral appliance in the mouth during sleep. The appliance covers the upper and lower teeth and acts to pull the lower jaw forward, opening the throat passage and allowing normal breathing.

Oral appliance treatment does not treat sleep apnea effectively in all patients. In order to identify those patients for whom oral appliance therapy will work, Zephyr Sleep Technologies has invented a remotely controlled device that tests various positions of the lower jaw. This commercially available device, known as MATRx, is an FDA-cleared motorized dental positioner that can be used in an overnight sleep study performed in the hospital or clinic. Temporary dental-impression trays cover the upper and lower teeth. These are attached to a small motor that slowly and gently pulls the lower jaw forward under the control of a technician who determines when the best position is reached. Knowing the best position, and the likelihood of future success, allows the dentist to build an oral appliance with confidence.

In order to eliminate the need for an overnight in-hospital sleep study, Zephyr Sleep Technologies has invented a new investigational device that allows clinicians to decide whether or not an individual is likely to benefit from oral appliance therapy, from the comfort of the individual's own home. An investigational device is one that is not cleared by the U.S. Food and Drug Administration (FDA). Like the MATRx, the patient sleeps with a motorized positioner that moves the lower jaw. However, the new device (called MATRx plus) is automatically controlled by a computer, rather than a sleep technician, making it a feedback controlled mandibular positioner. Participation in this study will provide important data regarding the use of these device in their intended commercial setting, the dentist's office.

Zephyr has previously carried out three research studies leading to the development of this feedback controlled mandibular positioner. The first study showed that the technician controlled positioner was able to accurately identify patients suitable for oral-appliance therapy, i.e., those with a good likelihood of success with a permanent device.

This study also identified the amount of jaw protrusion (how far forward the lower jaw needs to be pulled) that will provide therapeutic relief of the patients' sleep apnea. This trial resulted in the placement of the device on the market, now sold in the United States as MATRx. The second two trials showed that the feedback controlled software used by the new positioner was very accurate and was able to identify successful candidates in a home setting.

No serious or permanent problems or risks were identified in any of these research studies. Participants reported minor tooth and gum discomfort on the morning following the test and other minor issues including canker sores, excess saliva and being unable to sleep. Since other studies were designed to establish the safety and efficacy of the device, the purpose of the present research study is to collect additional data regarding the workflow of the device as it would occur during commercial use.

The test will occur over a series of nights in the home or during a single night in the sleep laboratory. The test type will be decided by the care providers and this study will only document the rationale and will not influence the choice of test. Participants will be asked to provide feedback as to the preferred test, and will be told if they are candidates for oral appliance therapy based on the output of the test.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Participant has been deemed suitable for oral appliance therapy
* Adequate mandibular range of motion
* Adequate dentition
* Ability to understand and provide informed consent
* Ability and willingness to meet the required schedule

Exclusion Criteria:

* Loose teeth or advanced periodontal disease
* Full dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of MATRx plus use in a dental sleep medicine practice, as determined by successful completion of test | 1 week
  Evaluation of the process to effectively coordinate the respective roles in the deployment of the sleep test. Feasibility will be determined by the ability for patients to complete the MATRx plus test.

SECONDARY OUTCOMES:
Patient satisfaction of test, as determined by feedback from the patients following the test. | 1 week
  Questionnaire on patient preference and feedback with respect to the test.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Moore, DDS, MD, Principal Investigator — Charlotte Oral Surgery
Locations (1):
- Charlotte Oral Surgery, Charlotte, North Carolina, United States